CLINICAL TRIAL: NCT03134664
Title: Supercapsular Percutaneously Assisted Total Hip Approach for the Elderly With Femoral Neck Fractures: a Prospective, Open-label, Randomized, Controlled Clinical Trial
Brief Title: Supercapsular Percutaneously Assisted Total Hip Approach for the Elderly With Femoral Neck Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Pudong Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShanghaiPudongH_002
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Femoral Neck Fractures
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Forty patients with femoral neck fractures admitted at Pudong Hospital of Fudan University, China are randomly divided into two groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients with femoral neck fractures are randomly assigned to undergo femoral head replacement via the SuperPATH approach in the experimental group.
  Interventions: Procedure: Experimental group
- Control group (Experimental): Patients with femoral neck fractures are randomly assigned to undergo femoral head replacement via the conventional posterior approach in the control group.
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: Experimental group — Patients with femoral neck fractures are randomly assigned to undergo femoral head replacement via the SuperPATH approach in the experimental group.
  Arms: Experimental group
Procedure: Control group — Patients with femoral neck fractures are randomly assigned to undergo femoral head replacement via the conventional posterior approach in the control group.
  Arms: Control group

SUMMARY:
To test that the SuperPATH approach is more safe and reliable for hip functional recovery compared with the postolateral approach in the artificial hip replacement for femoral neck fractures in the elderly.

DETAILED DESCRIPTION:
Femoral neck fracture is one of the most common diseases in the elderly. Artificial hip replacement is currently the preferred treatment for femoral neck fractures, and characterized by no presence of postoperative bone nonunion, femoral head necrosis and other complications, though longer operative time and larger surgical incision are unavoidable. Patients undergoing artificial hip replacement can recover weight-bearing walk early after surgery, making rehabilitation rapid, to avoid a variety of complications, such as bed rests. Hip replacement via posterolateral approach is generally used, but limited by large incision, cutting off the extortor, and postoperative hip dislocation.

The minimally invasive approach for hip replacement has the advantages of less blood loss and less trauma compared with conventional approaches. The supercapsular percutaneously-assisted total hip (SuperPATH) approach (Appendix 1) is consistent with the posterolateral approach in the anatomical landmark, preserving all the advantages of the posterior approach. Compared with the conventional approaches, the SuperPATH approach has no neurovascular interface that is uneasy to damage blood vessels and nerves during operation, reducing intraoperative blood loss, and retains all of the joint capsules and supinator muscles, significantly reducing the probability of postoperative dislocation of the hip. Osteotomy via this approach can be completed without hip dislocation, thus reducing incidence of vascular distortion and postoperative deep vein thrombosis. Hip replacement via the SuperPATH approach can be completed under direct vision rather than perspective inspection, and the surgical incision on the femur is made according to the femoral anteversion angle. In addition, this approach is also used for femoral intramedullary nail implantation. These surgical procedures are more likely to be grasped by clinicians. Preservation of the joint capsule and supinator muscles makes physical activities unrestricted and speeds up rehabilitation. Moreover, there is a corresponding reduction in the hospital stay and costs. However, SuperPATH technology is rarely reported in China as it has been introduced for a short time and in few hospitals.

Previous studies have reported that SuperPATH approach for artificial hip replacement exhibits better short-term effect on elderly femoral neck fractures. In this trial, the follow-up period will be prolonged to 6 months in order to observe the short-to-mid term effect in the elderly with femoral neck fractures.

Adverse events Postoperative adverse events including incision pain and infection, back muscle pain, spinal cord/nerve injury, length inequality of the lower limbs, prosthesis falling-off and prosthetic loosening will be recorded during the follow-up period. If severe adverse events occur, details including the data of occurrence, type of adverse events and therapeutic measures will be reported to the project manager and the institutional review board within 24 hours.

Data collection, management, analysis, and open access Data collection Clinical data, including demographic data, disease diagnosis, accompanying diseases, and allergic history (drug allergy), will be collected and summarized using standardized case report forms. These data will be processed and recorded electronically.

Data management Researchers will be responsible for data processing, confirming and locking. The locked data will be unable to be altered and preserved by the Pudong Hospital of Fudan University. In addition to these researchers, only the persons who have permission will have the right to query the database.

Data analysis All data will be statistically analyzed by professional statisticians who will responsible for completing an outcome analysis report that will be submitted to the principle investigator who will be responsible for completing a research report. An independent data monitoring committee is responsible for data monitoring and management throughout the entire trial to ensure scientific accuracy, stringency, authenticity, and integrity.

ELIGIBILITY:
Inclusion Criteria:

* Femoral head fractures as diagnosed by X-ran and CT;
* Garden III, IV;
* An age of > 75 years;
* Both genders.

Exclusion Criteria:

* Fractures with spinal cord injury;
* Fractures with nerve injury;
* Refusal to sign the informed consent.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Harris hip scores | changes of baseline, week 1 and month 6 postoperatively
  To assess hip function recovery in patients. The hip function is assessed by Harris scores ranging from 0-100: excellent ≥ 90, good 80-90, fair 70-79, bad < 70. The higher scores indicate better hip function.

SECONDARY OUTCOMES:
Length of surgical incision | during the surgery
  A smaller surgical incision causes smaller surgical trauma to patients.
Intraoperative blood loss | during the surgery
  Less blood loss indicates the surgical practice is more normative and safe.

CONTACTS AND LOCATIONS:
Overall Officials: Lianghao Wu, Ph.D, Principal Investigator — Pudong Hospital of Fudan University

IPD SHARING:
Plan to Share IPD: Undecided